CLINICAL TRIAL: NCT04447053
Title: Sequential Belimumab Followed by T-cell Based Therapy in the Treatment of Systemic Lupus Erythematosus (SUBTLE) - a Preliminary Proof-of-concept Mechanistic Study
Brief Title: Sequential Belimumab and T-cell Based Therapy in SLE
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National University Hospital, Singapore (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 10743-SUBTLE
Record Dates: First submitted 2020-06-23; First posted 2020-06-25 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Systemic Lupus Erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — belimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Belimumab + SOC (Experimental): Patients will be administered Belimumab, 10mg/kg, intravenously (IV) (together with SOC) in 1 hour on days 0, 14, and 28, and then every 28 days (4 weeks) until week 48.
  Interventions: Drug: Belimumab Injection [Benlysta]
- SOC only (No Intervention): Patients will receive SOC based on the discretion of attending physicians in accordance with the clinical disease manifestations of SLE and NUH practice of the treatment of SLE.

INTERVENTIONS:
Drug: Belimumab Injection [Benlysta] — Belimumab, IV infusion, 10mg/kg on days 0, 14, 28 then every 28 days until week 48.
  Arms: Belimumab + SOC

SUMMARY:
Systemic lupus erythematosus (SLE) is a disease in which the immune system (the bodily system that fights infection) attacks the body's own cells and tissues, causing inflammation and organ damage if not promptly and appropriately managed. Autoantibodies (specific proteins produced by the immune system which participate in attacking self tissues and organs) are the hallmarks of SLE which are produced by a specific type of white blood cells called B cells. Belimumab (Benlysta®) is a monoclonal antibody against the B cells by blocking the action of BLyS, a protein that prolongs the longevity and enhances the functions of B cells and is found to be elevated in patients with SLE, was approved by the FDA to treat patients with SLE. This study aims to study the effects of Belimumab on T cells, another specific type of white blood cells which also play a crucial role in SLE, in patients with SLE. In this trial, 80 adult patients with SLE will be recruited, 40 of them will be assigned to receive intravenous (IV) Belimumab with standard of care therapy (SOC), and 40 to receive SOC only. After 48 weeks of exposure to Belimumab + SOC and SOC alone, the phenotype and functions of T cells will be studied and compared.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 21
2. Able to understand the details of the trial and willing to give written informed consent and comply with the requirements of the study protocol.
3. Patients who fulfill the classification criteria (SLICC 2012 or ACR 1997) for SLE and have active disease (SELENA-SLEDAI ≥ 6).
4. Patients whose sera are positive for ANA (titre ≥ 1:80) or anti-dsDNA (>100U/L based on NUH standard laboratory cut-off).
5. Patients who are on stable dose of prednisolone (0-40mg/day) and/or non-steroidal anti-inflammatory, antimalarial or immunosuppressive drugs for at least 30 days before first study dose.
6. Females of child-bearing potential and non-sterilized males with female partners of child-bearing potential may participate this trial only if they use a reliable means of contraception.
7. Females of child-bearing potential must have a negative serum pregnancy test within three weeks prior to baseline.

Exclusion Criteria:

1. They have severe active nephritis and/or active CNS lupus and/or other autoimmune diseases e.g. RA, mixed connective tissue disease, scleroderma, dermatomyositis and polymyositis.
2. They are pregnant.
3. They have had previous treatment with any B-cell and T-cell targeted biologic therapy, intravenous (IV) cyclophosphamide within 6 months of enrolment, intravenous immunoglobulins or prednisolone (>100mg/day) within 3 months.

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-11-08 (Actual); Primary Completion 2025-05-20 (Estimated); Study Completion 2025-05-20 (Estimated)

PRIMARY OUTCOMES:
Comparing the ratio of Treg/Teff in Belimumab + SOC arm with SOC-only arm | Baseline, week 4, week 12, week 24, week 36, week 48 and week 60
  The enumeration of T-cell subsets by multi-color flow cytometry including Th1 (CD4+Tbet+), Th2 (CD4+GATA3+), Th17 (CD4+RoRgamat+) and Treg (CD4+CD25+FoxP3+) cells, as well as CD19+CD20+ B cells after staining with respective fluorescent-conjugated antibodies.
Identifying and comparing the TCR sequence of the variable regions (CDR1, CDR2 and CDR3) and their RNA expression profile before and after 48 weeks of Belimumab therapy | up to week 48
  TCR sequencing and RNA expression with the use of the state-of-the-art 10x Genomic nano-droplet technology.

SECONDARY OUTCOMES:
To compare the numeric difference in other T cell subsets (Th1, Th2 and Th17) between the 2 arms | Baseline, week 4, week 12, week 24, week 36, week 48 and week 60
  The enumeration of T-cell subsets by multi-color flow cytometry.
To compare the potential improvement of cognitive function between the 2 arms | Baseline and week 52
  The use of the computerized Automated Neuropsychological Assessment Matrix (ANAM) which serves as an initial screening tool to pick up subtle cognitive dysfunction in healthy populations and serial assessments to track the progress of cognitive dysfunction in SLE patients over time.

CONTACTS AND LOCATIONS:
Overall Officials: Anselm Mak, Principal Investigator — National University Hospital, Singapore
Locations (1):
- National University Hospital, Singapore, Singapore